CLINICAL TRIAL: NCT01363609
Title: Central Effects of Endogenous Glucagon Like Peptide-1 (GLP-1) and the GLP-1 Analog Liraglutide on Brain Satiety and Reward Circuits and Feeding Behavior in Diabetes
Brief Title: Effects of Glucagon Like Peptide-1(GLP-1) and Liraglutide on Brain Satiety and Reward Circuits and Feeding Behavior in Diabetes
Acronym: LIBRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, RG IJzerman, MD, PhD, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: DC2011LiBrain001
Record Dates: First submitted 2011-05-26; First posted 2011-06-01 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Obesity; Type 2 Diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Liraglutide (Experimental): 12 week treatment with liraglutide in fixed dosage
  Interventions: Drug: Liraglutide treatment 12 weeks
- Insulin glargine (Active Comparator): 12 week treatment, once daily, with insulin glargine. Dosage based on fasting blood glucose measurements
  Interventions: Drug: insulin glargine treatment
- before start of treatment period (Other): before start of the treatment period, one day with tests will be performed. During this test a GLP-1 receptor antagonist will be administered In the group with obesity and planned gastric bypass surgery, the GLP-1 receptor agonist will be administered during 1 test before and 1 test after the surgery
  Interventions: Drug: GLP-1 receptor antagonist

INTERVENTIONS:
Drug: Liraglutide treatment 12 weeks — liraglutide will be started with a titration period of 2 weeks: week 1 0.6mg once daily, week 2 1.2mg once daily. If well tolerated, treatment will be continued for 10 more weeks in dosage of 1.8mg once daily
  Arms: Liraglutide
Drug: insulin glargine treatment — Insulin glargine treatment consist a treatment period of 12 weeks. Treatment will start with a dosage of 10 IU once daily. Patient will self-titrate the insulin glargine dosage based on self-monitored fasting blood glucose (FBG) concentrations for the previous 3 days using the following guideline: If FBG levels are above 5.6 mmol/L (100-153 mg/dL) on 3 consecutive mornings, the daily dose is to be increased by 2 IU/day. If hypoglycemia documented by glucose concentration < 3.3 mmol/L (60 mg/dL) or requiring assistance occurs without an easily identifiable reason (skipped meal, excessive physical activity), the daily dose is to be downregulated, with -2 IU/day
  Arms: Insulin glargine
Drug: GLP-1 receptor antagonist — Exendin 9-39 will be infused intravenously at doses of 600 pM/kg • min. This will only be during one of the visit for the healthy lean controls and the T2DM group, and during two visits in the group with obesity planned for gastric bypass surgery
  Arms: before start of treatment period

SUMMARY:
The aim of this study is to investigate if endogenous Glucagon Like Peptide -1 (GLP-1) has an effect on brain satiety and reward systems and if there are alterations in obese patients with type 2 diabetes (T2DM). Secondly, the aim is to investigate whether treatment with a GLP-1 analog, liraglutide, restores these signals in obese patients with type 2 diabetes. Finally, also the endogenous GLP-1 effects will be investigated in obese individuals before and after gastric bypass surgery on brain satiety and reward systems.

DETAILED DESCRIPTION:
First aim will be addressed in a cross-sectional randomized study. 20 healthy, lean and 20 obese individuals with type 2 diabetes (T2DM) will be exposed to food cues and with concomitant infusion of glucagon Like peptide-1 (GLP-1) receptor antagonist or saline, to assess the involvement of endogenous GLP-1, secreted in response to a meal. Measurements activation of CNS circuits involved in satiety and reward will be performed using blood oxygen level-dependent (BOLD) functional magnetic resonance imaging (fMRI).

The second aim will be addressed in cross-over randomized-controlled trial (RCT) in the T2DM patients only. Patients will be randomly assigned liraglutide vs insulin glargine treatment, during a treatment period of 12 weeks each with a 12-week washout period in between. The investigators will perform the same fMRI protocol.

The third aim will be addressed in a study with obese individuals who are scheduled for a gastric bypass surgery. The same protocol as for the first aim will be performed and this will be before and after the surgery in the same individuals.

ELIGIBILITY:
Inclusion Criteria:

* For the healthy, lean individuals:
* Age 18-65 years
* Women: post menopausal (excluding possible menstruation cycle effects)
* Body-mass index (BMI) of <25 kg/m2,
* Stable bodyweight (<5% reported change during the previous 3 months).
* Normal fasting and 2h post load glucose as ascertained during a 75-g oral glucose tolerance test (OGTT) (34)
* Right handed

For the obese T2DM individuals:

* Age 18-65 years
* Women: post menopausal (excluding possible menstruation cycle effects)
* BMI 25-40 kg/m2
* Stable bodyweight (<5% reported change during the previous 3 months).
* Diagnosed with T2DM > 3 months prior to screening
* HbA1C 6.5-8.5%
* Treatment with metformin at a stable dose for at least 3 months.
* Right handed

For the obese individuals scheduled for gastric bypass surgery:

* Age 18-65 years
* Women: preferably post menopausal (excluding possible menstruation cycle effects)
* Body-mass index (BMI) of >30 kg/m2,
* Stable bodyweight (<5% reported change during the previous 1 months).
* Normal or impaired fasting and 2h post load glucose as ascertained during a 75-g oral glucose tolerance test (OGTT) (defined as glucose fasting < 7.1 mmol/l and after OGTT t=120min < 11.0 mmol/l) (39)
* Right handed

Exclusion Criteria:

* GLP-1 based therapies, thiazolidinediones, sulphonylurea or insulin within 3 months before screening
* Weight-lowering agents within 3 months before screening.
* Congestive heart failure (NYHA II-IV)
* Chronic renal failure (glomerular filtration rate < 60 mL/min/1.73m2 per Modification of Diet in Renal Disease (MDRD))
* Liver disease
* History of gastrointestinal disorders (including gastropareses, pancreatitis and cholelithiasis)
* Neurological illness
* Malignancy
* Other type of bariatric surgery (Redo-GBP, sleeve, distal GBP, adj banding, Scopinaro)
* History of major heart disease
* History of major renal disease
* Pregnancy or breast feeding
* Implantable devices
* Substance abuse
* Addiction
* Contra-indication for MRI, such as claustrophobia or pacemaker
* Any psychiatric illness; including eating disorders and depression
* Chronic use of centrally acting agents or glucocorticoids within 2 weeks immediately prior to screening.
* Use of cytostatic or immune modulatory agents
* History or known allergy for acetaminophen.
* History of allergy for insulin analog
* History of allergy for liraglutide
* Participation in other studies
* Individuals who have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry
* Individuals who are investigator site personnel, directly affiliated with the study, or are immediate family

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
food-stimuli related neuronal activity in reward and satiety circuits as represented by BOLD fMRI signal change from baseline (%) | approximately 3 years
  * differences between obese T2DM patients and healthy lean subjects food-stimuli related neuronal activity in reward and satiety circuits as represented by BOLD fMRI signal change from baseline (%)
  * the involvement of endogenous GLP-1 food-stimuli related neuronal activity in reward and satiety circuits as represented by BOLD fMRI signal change from baseline (%)
  * Effects of treatment with the GLP-1 analog liraglutide in obese patients with type 2 diabetes in food-stimuli related neuronal activity in reward and satiety circuits as represented by BOLD fMRI signal change from baseline (%)
  * - To investigate the involvement of the increased meal-related endogenous GLP-1 levels after gastric bypass surgery in these food-stimuli related CNS satiety and reward responses and to investigate whether pharmacological blocking of endogenous GLP-1 receptor activation, using a GLP-1 antagonist, differentially affects these responses before and after gastric bypass surgery in obese individuals.

SECONDARY OUTCOMES:
GLP-1 analog treatment related changes in obese patients with type 2 diabetes in self-reported hunger, satiety, fullness | approximately 3 years
GLP-1 analog treatment related changes in obese patients with type 2 diabetes in basal metabolic rate and post-prandial energy expenditure | approximately 3 years
GLP-1 analog treatment related changes in obese patients with type 2 diabetes in microvascular function and vasomotion | approximately 3 years
GLP-1 analog treatment related changes in obese patients with type 2 diabetes in cardiovascular autonomic nervous balance | approximately 3 years
GLP-1 analog treatment related changes in obese patients with type 2 diabetes in concomitant changes in metabolic and humoral markers | approximately 3 years
Alterations in resting state brain activity networks in obese patients with type 2 diabetes compared to lean, healthy individuals and the involvement of endogenous GLP-1 | approximately 3 years
Alterations in brain arterial blood flow in obese patients with type 2 diabetes compared to lean, healthy individuals and the involvement of endogenous GLP-1 | approximately 3 years
GLP-1 analog treatment related changes in obese patients with type 2 diabetes in resting state brain activity networks. | approximately 3 years
GLP-1 analog treatment related changes in obese patients with type 2 diabetes in brain arterial blood flow. | approximately 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- VU University Medical Center, Amsterdam, Netherlands

REFERENCES:
- [Derived] Ten Kulve JS, Veltman DJ, Gerdes VEA, van Bloemendaal L, Barkhof F, Deacon CF, Holst JJ, Drent ML, Diamant M, IJzerman RG. Elevated Postoperative Endogenous GLP-1 Levels Mediate Effects of Roux-en-Y Gastric Bypass on Neural Responsivity to Food Cues. Diabetes Care. 2017 Nov;40(11):1522-1529. doi: 10.2337/dc16-2113. PMID 29025878
- [Derived] ten Kulve JS, Veltman DJ, van Bloemendaal L, Barkhof F, Deacon CF, Holst JJ, Konrad RJ, Sloan JH, Drent ML, Diamant M, IJzerman RG. Endogenous GLP-1 mediates postprandial reductions in activation in central reward and satiety areas in patients with type 2 diabetes. Diabetologia. 2015 Dec;58(12):2688-98. doi: 10.1007/s00125-015-3754-x. Epub 2015 Sep 18. PMID 26385462